CLINICAL TRIAL: NCT01774539
Title: Diffusion MRI as a Prognostic Tool in Growth Plate Injuries: A Pilot Study to Assess Feasibility
Brief Title: Diffusion MRI and Growth Plate Injuries: Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Pediatric Orthopaedic Society of North America (Other)
Responsible Party: Sponsor
Other Study IDs: H12-03016
Record Dates: First submitted 2013-01-22; First posted 2013-01-24 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Fracture
Keywords: Fracture; Physeal injury; Diffusion MRI
MeSH Terms: conditions — Fractures, Bone | interventions — Diffusion Tensor Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Physeal Injury - Distal Radius: Patients who suffer a physeal fracture of the distal radius will be scanned and compared to their healthy contralateral limb.
  Interventions: Other: Diffusion MRI

INTERVENTIONS:
Other: Diffusion MRI — Each subject will undergo one diffusion MRI scan to identify characteristics of their physes

SUMMARY:
Children who suffer fractures to the growth plates (physes) of their bones are at risk for premature growth arrest which can lead to long term complications. There is currently no technique to predict who is at risk of growth arrest following a physeal injury. The investigators aim to determine if diffusion MRI (an imaging method to analyze tissue properties) can effectively pick up differences between a healthy growth plate and an injured one. This would allow orthopaedics surgeons to predict which injuries are at a higher risk of growth arrest, so earlier interventions can be done in the orthopaedic clinic.

DETAILED DESCRIPTION:
The purpose of this study is to determine if diffusion MRI can be used for tissue characterization in childhood and adolescent growth plate injuries, and to get a better understanding of the physiologic disturbance of an injured physis

ELIGIBILITY:
Inclusion Criteria:

* Salter-Harris Type II, III, or IV fracture through the distal radius
* Growth plates are open
* Ages 8-12
* Able to consent in English

Exclusion Criteria:

* All fractures not sustained to distal radius
* SH Type I or V fracture
* Injury to contralateral limb
* Previous injury to distal radius
* Diseases known to alter bone healing or growth]
* Contraindications to undergoing an MRI scan

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Study subjects will be selected from the Orthopaedic Trauma Clinic at BC Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Tissue characterization of growth plate using diffusion MRI | 4-6 weeks following injury
  Diffusion MRI scan of injured and contralateral (control) physis.

CONTACTS AND LOCATIONS:
Overall Officials: Firoz Miyanji, MD, FRCSC, Principal Investigator — University of British Columbia
Locations (1):
- British Columbia Children's Hospital, Vancouver, British Columbia, Canada